CLINICAL TRIAL: NCT03625817
Title: A Randomized Cross Over Trial About the Influence of Skin Temperature Gradient on the Variation of Metabolic Hormones in Climates With Different Ambient Air Temperatures
Brief Title: Skin Temperature Gradient Effects on the Variation of Metabolic Hormones in Adults
Acronym: TEMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Konstantinos Makris, Dean and Associate Professor of Environmental Health at School of Health Sciences, Director of Water and Health Lab, Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CUT2
Record Dates: First submitted 2018-07-13; First posted 2018-08-10 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Temperature Change, Body; Stress; Metabolic Disturbance
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: A 2 x 2 cross-over pilot study of healthy adults is proposed to prospectively describe the effect of ambient temperature gradient on metabolic hormonal secretion patterns. A total of 50-60 subjects will be followed for a period of 7 days firstly in an urban environment or in a village of the mountainous rural environment and later, for the same period, in the alternate setting, during the summer period in Cyprus. The two settings will allow for the comparison of the circadian patterns of hormones secreted by the adipose tissue among different gradient temperature changes. Continuous quantification of skin temperatures on one day in each setting will allow for characterization of how skin temperature is affected by ambient temperature. Collection of all urine voids in one day in each setting will allow for quantification of the hormone secretion by the adipose tissue.
Who Masked: Investigator, Outcomes Assessor
Masking Description: There will be the necessary blinding during the conduct of the all laboratory and statistical analyses. At the start of the study, participants will be given a 2-digit code (10-60) - once the researchers have names of eligible participants, each name will be given a code. This will be participant's study ID that will accompany participant's answered questionnaires, diaries, urine vials and temperature measurement's files.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban setting (No Intervention): The participants will be staying in their permanent house in an urban area in Cyprus for at least 7 days. On the 7th day, they will be wearing 2 temperature sensors, for skin and air temperature. They will also collect the urine samples of the day and note in an activity diary, the names and times of activities.
- Mountainous setting (Experimental): The intervention is the short stay in the mountainous area of Troodos for atleast 7 consecutive days. The participants will be staying in their holiday house in the mountainous-rural area of Troodos, Cyprus for at least 7 days. On the 7th day, they will wear 2 temperature sensors, for skin and personal air temperature monitoring (every minute data points). They will also collect the urine samples of the day and note in an activity diary, the names and times of activities.
  Interventions: Behavioral: Mountainous setting

INTERVENTIONS:
Behavioral: Mountainous setting — The mountainous setting is characterized by lower temperatures (about 8-10C ambient air temp.) than those in urban setting, also having >800m altitude.Each period will last for 1 week with a wash out period of minimum 2 days. Continuous skin temperature and ambient temperature monitoring will take place in the last day of each period, towards the end. During the 2 sampling days, 24-hour urine voids will be collected in different vials. Participants will be required to fulfill a diary with their daily activities, meal times, collection of urine times, sleep/wake times and times of leaving/entering a closed environment.
  Arms: Mountainous setting

SUMMARY:
The Cyprus International Institute for Environmental and Public Health of the Cyprus University of Technology is planning a pilot study of health indicators in relation to spatially varying climatic conditions ranging from the city to the mountainous environment. The purpose of the project is to understand the effect of fluctuations in external climatic conditions on the human body temperature and metabolic biomarkers or stress hormones.

Climate change phenomena such as protracted heat waves that create areas with even higher temperatures, especially in urban centers, may have a negative impact on human health. The effects may be acute for an individual with the appearance of discomfort and headaches, while chronic exposures to high air temperatures for the general population have been linked with premature mortality and cardiovascular diseases. Due to climate change that is hitting hard the Mediterranean, these temperature changes have been more and more common in Cyprus in recent years.

One of the usual ways of dealing with high temperatures is the use of air conditioners. With sudden and frequent temperature changes during the day, the human body is subject to thermal shock for varying duration and number of times, having wear and tear consequences for the human physiology. The investigators hypothesized that the number, duration and frequency of human exposures to wide gradient (> 8 ° C) of air temperature changes may be related to potential health problems. An intervention potentially reducing the health risk associated with extended exposure to high temperatures in the summer for Cypriots may be the temporary (for a few days or hours) stay in the villages of mountainous area. Most of the mountain communities in Cyprus have consistently lower mean ambient air temperatures of about 10 degrees Celsius than those in the cities, so the investigators anticipate not observing the metabolic hormone alterations induced while being in the city environment.

DETAILED DESCRIPTION:
A randomised crossover trial study design was used to: investigate the circadian patterns of metabolic adipokines (leptin, adiponectin and ghrelin hormones), using targeted biomarker measurements and untargeted metabolomics in healthy adults residing in two different climatological environments: urban and higher in latitude mountainous settings, and ii) investigate the effect of skin temperature gradient on the variation of adipokines in the two settings (urban and rural).

The study will take place in Cyprus. Participant recruitment will abide by the ethical principles and the guidelines of the National Bioethics Committee of Cyprus. Participants will be recruited after they read and complete the consent form and the whole study protocol is explained to them. Information about the study will be disseminated through flyers and through telephone communication via governmental and other non-profitable organizations that will contact community leaders of the area and help us collect and create a contact list of "Potential Participants". From there, potential participants will be informed about the study and screened for eligibility criteria via telephone.

Upon consent, the "Potential Participants List" will have to be randomized to assign the participants in to two different groups. A total of 50-60 subjects will be followed for a period of one week firstly in an urban environment and later, for the same period, in a village of the mountainous rural environment, during the summer period in Cyprus.

Once the researchers have names of potential participants, each name will be given a 2-digit code. This will be participant's study ID that will accompany participants answered questionnaires, diaries, urine vials and temperature measurement's files. The preparation of each tool with filled participants ID code and Date will be made at priory.

There will be no blinding since the interventions are known to the participants and the researchers. There will be the necessary blinding during the conduct of the all laboratory and statistical analyses.

The field workers and participants will arrange four visits. Visit 1 and 3 will take place one day before the sampling day which is the last day at each site(urban Vs rural), whereas visit 2 and 4 will take place a day after the sampling day when collection of the data will take place.

Except the preparation for the first sampling day during the first visit, participants will be asked to sign the informed consent form and to fill in two survey questionnaires (baseline characteristics and chronotype questionnaire). During sampling days, participants will be handed with the diary of activities, urine vials for urine sample collection and the instructions form (for urine collection and the use of the personal temperature sensors). Electronic temperature sensors should be activated by the researchers on the spot and placed on the participant during the first and third visit. The temperature data collection will be ensured on the spot during the second and forth visit. Participants will be asked to collect urine voids by collecting all bladder content during urination in vials provided by the Water and Health Lab. The first urine void of each sampling day will be discarded. All urine voids for the rest of the sampling day, of each participant, will be collected, including the first urine void of the following day. Samples will be kept at a freezer by the participant until collected by a member of the research team, in cool boxes. Upon arrival at the Water and Health lab samples, aliquoting will take place and then aliquot samples will be stored in freezers of -80◦C, until analysis.

Data collected will be digitized, anonymized and statistically evaluated. All data management steps will be employed to ensure that a final, clean, tidy and replicable dataset will be produced before proceeding to the statistical analysis. Descriptive statistics of the study population will be performed that will include parameters such as the mean and standard deviation for continuous variables and percentages for variables that indicate proportions.

The effect of temperature gradient changes and hormonal level, as well as, differences in cortisol levels between and within subject variation will be examined. The statistical analyses will include a range of approaches from descriptive statistics to regression analysis and metabolomics analyses. Pre-post analyses, non-linear mixed effects models, will be used to identify correlations of the circadian rhythms of the participants between the two settings. Statistical evaluation and graphical presentation of results will be prepared for a final report and presentation. All statistical analyses will be conducted at the Water and Health laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 20-60 years old
* Those that intend staying in mountainous area of Cyprus for the period of at least 1 week between July and September 2018

Exclusion Criteria:

* Pregnant women
* Obese individuals (>30 kg m-2)
* Those that have travelled to another country within one week of the study start date.
* People with history of hypertension or with diabetes or metabolic syndrome, or cancer.
* People receiving pharmaceutical treatment for impaired glucose levels and/or hypertension and/or antidepressants or thyroxin for thyroid disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline for adipokines (leptin, adiponectin and ghrelin) at day seven | units of measure are the same for all these hormones as ng/g. 1 day in the mountainous setting and 1 day in the urban setting (three spot urine samples per day per participant)
  First morning, and last before sleep of urinary adipokines measured with immunoassay kits
Change from baseline for stress hormones (melatonin and cortisol) at day seven | units of measure for all these hormones as ng/g. 1 day in the mountainous setting and 1 day in the urban setting (three spot urine samples per day per participant)
  First morning, last before sleep of cortisol/melatonin measured in urine with mass spectrometry

SECONDARY OUTCOMES:
Metabolite differences | these will have the same units of measure as ug/g. 1 day in the mountainous setting and 1 day in the urban setting
  Differentiated metabolite change (fold change) for metabolomics platform-based profiles of in two study settings with distinctly different climatological characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos C Makris, PhD, Principal Investigator — Cyprus International Institute of Environmental and Public Health
Locations (1):
- Cyprus International Institute of Environmental and Public Health, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
Urine Analysis data of the individual are to be saved and used for future research, after participants' consent.

REFERENCES:
- [Derived] Makris KC, Charisiadis P, Delplancke T, Efthymiou N, Giuliani A. Diurnal Nonlinear Recurrence Metrics of Skin Temperature and Their Association with Metabolic Hormones in Contrasting Climate Settings: A Randomized Cross-Over Trial. Int J Environ Res Public Health. 2022 Nov 17;19(22):15195. doi: 10.3390/ijerph192215195. PMID 36429912

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03625817/SAP_000.pdf